CLINICAL TRIAL: NCT04896762
Title: Extrapulmonary Presentation of COVID-19 Patients During the Second Wave
Brief Title: Extrapulmonary Presentations of COVID-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hend Mohammed Abdelraheem Esmaeel, assistant professor, Sohag University
Other Study IDs: Soh-Med-21-04-25
Record Dates: First submitted 2021-05-15; First posted 2021-05-21 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
Keywords: extrapulmonary presentation; pulmonary
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Extrapulmonary presentation for COVID-19: patients with confirmed covid 19 disease who primarily presented with extrapulmonary system affection
- pulmonary presentation for COVID-19: patients with confirmed covid 19 disease who primarily presented with pulmonary disease

SUMMARY:
An observational study about the extrapulmonary presentations of COVID-19 patients during the second wave of the pandemic.

DETAILED DESCRIPTION:
a prospective observational study that aimed at

1. provide an overview about the prevalence of extra-pulmonary presentation of COVID-19 during the second wave of the pandemic and
2. Detection of the most frequent affected systems with comparison between the pulmonary and extrapulmonary presentation of COVID 19 as regard patient demographics, comorbidity and level of care needed.

ELIGIBILITY:
Inclusion Criteria:

* all patient with confirmed covid 19 disease presented to our health facility during the second wave of the pandemic

Exclusion Criteria:

* other diagnosis than covid 19 as a primary cause of presentation of the patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients presented at a triage point in a tertiary health care facility with a suspected covid 19 disease.
Sampling Method: Probability Sample
Enrollment: 948 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
extrapulmonary presentation in COVID-19 | Baseline presentation of confirmed cases with COVID-19
  frequency of extrapulmonary presentation inCOVID-19 second wave pandemic

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dong E, Du H, Gardner L. An interactive web-based dashboard to track COVID-19 in real time. Lancet Infect Dis. 2020 May;20(5):533-534. doi: 10.1016/S1473-3099(20)30120-1. Epub 2020 Feb 19. No abstract available. PMID 32087114
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013